CLINICAL TRIAL: NCT01193946
Title: Assessment of Dietary Protein Needs of Older Women
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Other Study IDs: 1001008857; UL1RR025761 (NIH)
Record Dates: First submitted 2010-07-27; First posted 2010-09-02 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Protein-energy; Imbalance
Keywords: Protein requirement; Elderly women; Indicator amino acid oxidation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single-arm design: There is currently considerable debate regarding the accuracy of the estimated average requirement (EAR) and the recommended dietary allowance (RDA) for older people. Very limited data obtained from older individuals are available to support the assumption that age does not affect protein requirement. Existing method like nitrogen balance has inherent limitations that diminish it from being considered a reference method. Indicator amino acid oxidation technique is emerging as an alternative method to measure dietary protein requirement. It is more accurate and less demanding. The current study will be the first time this technique is used with elderly adults and will provide an important foundation for geriatric nutrition research
  Interventions: Dietary Supplement: dietary control

INTERVENTIONS:
Dietary Supplement: dietary control — Seven dietary protein levels will be tested randomly on the 7 testing days: 0.10, 0.30, 0.60, 0.90, 1.2, 1.5, and 1.8 g∙kg-1∙d-1.

SUMMARY:
The purpose of this study is to evaluate dietary protein requirements in elderly women aged 80 years and older using the indicator amino acid oxidation technique.

Hypothesis to be tested: Protein requirement for elderly women is higher than the estimated average requirement of 0.66 g∙kg-1∙d-1 protein. The recommended protein intake for elderly women is higher than the recommended dietary allowance of 0.80 g∙kg-1∙d-1 protein.

DETAILED DESCRIPTION:
There is currently considerable debate regarding the accuracy of the estimated average requirement (EAR) and the recommended dietary allowance (RDA) for older people. Very limited data obtained from older individuals are available to support the assumption that age does not affect protein requirement. Existing method like nitrogen balance has inherent limitations that diminish it from being considered a reference method. Indicator amino acid oxidation technique is emerging as an alternative method to measure dietary protein requirement. It is more accurate and less demanding. The current study will be the first time this technique is used with elderly adults and will provide an important foundation for geriatric nutrition research.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age range: 80 yrs and older
* Body mass index between 22-30
* Weight stable 4.5 kg weight gain or loss within the last 6 month
* Non-smoking within the last 6 month
* Ambulatory
* Clinically normal blood profiles within 10% of clinical normalc.
* No diseases or not taking medications known to influence protein or energy metabolism,
* Willingness and ability to consume food provided and not allergic to phenylalanine
* Continent, strong bladder control

Exclusion Criteria:

* Male,
* Gained or lost more than 4.5 kg of body weight within the last 6 months,
* Non-ambulatory (i.e. bedridden, wheel-chair bound),
* Clinically abnormal blood profiles as identified by our study physician, Arthur Rosen, MD

Min Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Female Age range: 80 yrs and older Body mass index between 22-30 Weight stable 4.5 kg weight gain or loss within the last 6 month Non-smoking within the last 6 month Ambulatory Clinically normal blood profiles within 10% of clinical normalcy. No diseases or not taking medications known to influence protein or energy metabolism, Willingness and ability to consume food provided and not allergic to phenylalanine
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
dietary protein requirement in older women | 3 month
  Dietary protein requirement is assessed by the subjects' differential response to different dietary protein intake

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Tang M, McCabe GP, Elango R, Pencharz PB, Ball RO, Campbell WW. Assessment of protein requirement in octogenarian women with use of the indicator amino acid oxidation technique. Am J Clin Nutr. 2014 Apr;99(4):891-8. doi: 10.3945/ajcn.112.042325. Epub 2014 Jan 15. PMID 24429540